CLINICAL TRIAL: NCT03674957
Title: The Manitoba Personalized Lifestyle Research (TMPLR) Study
Status: Terminated | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Research Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: HS18951(H2015:367)
Record Dates: First submitted 2018-04-12; First posted 2018-09-18 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2018-11

CONDITIONS: Diabetes; Cardiovascular Diseases; Chronic Kidney Diseases
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood (plasma, serum, red blood cells, white blood cells) samples, fecal samples, urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lifestyle factors, such as diet, physical activity and sleep, are associated with the development of many chronic diseases. The objective of The Manitoba Personalized Lifestyle Research (TMPLR) study is to understand how these lifestyle factors interact with each other and additional factors, such as an individual's genetics and gut microbiome, to influence health. This is an exploratory cross-sectional observational cohort study of adults, with extensive phenotyping by objective health and lifestyle assessments, and retrospective assessment of early life experiences, with retrospective and prospective utilization of secondary data from administrative health records. A planned non-random convenience sample of 840 Manitobans aged 30-46 recruited from the general population, stratified by sex (equal males and females), body mass index (BMI; 60% of participants with a BMI >25 kg/m2), and geography (25% from rural areas,). These stratifications were selected based on Manitoba demographics. Body composition and bone density will be measured by dual energy x-ray absorptiometry. Blood pressure, pulse wave velocity, and augmentation index will be measured on two consecutive days. Chronic disease risk biomarkers will be measured in blood and urine samples. DNA will be extracted for genetic analysis. A fecal sample will be collected for microbiome analysis.

DETAILED DESCRIPTION:
Lifestyle factors, such as diet, physical activity and sleep, are associated with the development of many chronic diseases. The objective of The Manitoba Personalized Lifestyle Research (TMPLR) study is to understand how these lifestyle factors interact with each other and additional factors, such as an individual's genetics and gut microbiome, to influence health. This is an exploratory cross-sectional observational cohort study of adults, with extensive phenotyping by objective health and lifestyle assessments, and retrospective assessment of early life experiences, with retrospective and prospective utilization of secondary data from administrative health records. A planned non-random convenience sample of 840 Manitobans aged 30-46 recruited from the general population, stratified by sex (equal males and females), body mass index (BMI; 60% of participants with a BMI >25 kg/m2), and geography (25% from rural areas,). These stratifications were selected based on Manitoba demographics. Lifestyle factors assessed will include dietary pattern, physical activity, cardiovascular fitness and sleep. Additional factors such as medical history, socio-economic status, alcohol and tobacco consumption, cognition, stress and anxiety, and early life experiences will also be documented. A maternal survey will be performed. Body composition and bone density will be measured by dual energy x-ray absorptiometry. Blood pressure, pulse wave velocity, and augmentation index will be measured on two consecutive days. Chronic disease risk biomarkers will be measured in blood and urine samples. DNA will be extracted for genetic analysis. A fecal sample will be collected for microbiome analysis. Participants may provide their Manitoba Personal Health Information Number (PHIN) to link their study data with administrative health records.Lifestyle factors, such as diet, physical activity and sleep, are associated with the development of many chronic diseases. The objective of The Manitoba Personalized Lifestyle Research (TMPLR) study is to understand how these lifestyle factors interact with each other and additional factors, such as an individual's genetics and gut microbiome, to influence health. This is an exploratory cross-sectional observational cohort study of adults, with extensive phenotyping by objective health and lifestyle assessments, and retrospective assessment of early life experiences, with retrospective and prospective utilization of secondary data from administrative health records. A planned non-random convenience sample of 840 Manitobans aged 30-46 recruited from the general population, stratified by sex (equal males and females), body mass index (BMI; 60% of participants with a BMI >25 kg/m2), and geography (25% from rural areas,). These stratifications were selected based on Manitoba demographics. Lifestyle factors assessed will include dietary pattern, physical activity, cardiovascular fitness and sleep. Additional factors such as medical history, socio-economic status, alcohol and tobacco consumption, cognition, stress and anxiety, and early life experiences will also be documented. A maternal survey will be performed. Body composition and bone density will be measured by dual energy x-ray absorptiometry. Blood pressure, pulse wave velocity, and augmentation index will be measured on two consecutive days. Chronic disease risk biomarkers will be measured in blood and urine samples. DNA will be extracted for genetic analysis. A fecal sample will be collected for microbiome analysis. Participants may provide their Manitoba Personal Health Information Number (PHIN) to link their study data with administrative health records.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have lived in Manitoba for a minimum of 5 years

Exclusion Criteria:

* Women who are pregnant or lactating are not eligible to participate

Ages: 30 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A sample of 800 Manitobans aged 30-46, stratified by sex, BMI, and geography are being recruited. Participants must have lived in Manitoba for a minimum of 5 years. Women who are pregnant or lactating are not eligible to participate. Additionally, because it is expected that very few of the 800 Manitobans who join TMPLR study from the general public will have reduced kidney function (eGFR <30 ml/min), 40 participants (20 female, 20 male, with no set stratification based on BMI or geography) who have severely reduced kidney function are being recruited from the renal health clinic at Seven Oaks General Hospital (Winnipeg, Manitoba).
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Percent fat mass | Baseline
  Measured using dual-energy X-ray absorptiometry
Percent lean mass | Baseline
  Measured using dual-energy X-ray absorptiometry
Bone mineral density | Baseline
  Measured using dual-energy X-ray absorptiometry, calculated as (mg/cm^2)

SECONDARY OUTCOMES:
(ASA24) dietary assessment tool | Baseline
  (ASA24) dietary assessment tool
Food energy intake | Baseline
  Assessed using dietary history questionnaire
Macronutrient intake | Baseline
  Assessed using dietary history questionnaire
Micronutrient intake | Baseline
  Assessed using dietary history questionnaire
Dietary restraint | Baseline
  Score 0-20 from Three-Factor Eating Questionnaire
Dietary disinhibition | Baseline
  Score 0-16 from Three-Factor Eating Questionnaire
Hunger | Baseline
  Score 0-14 from Three-Factor Eating Questionnaire
Pittsburgh sleep quality index | Baseline
  Pittsburgh sleep quality index
Montreal cognitive assessment questionnaire | Baseline
  Total score of 30; minimum score 0; maximum score of 30
Frailty status, as determined by the Modified Fried Criteria | Baseline
  Patients meeting the criteria for ≥ 3 of the following 7 criteria are deemed frail.
  1. Slowness - After two trials of a 5 m walk, average time>6 s
  2. Weakness - After three grip strength measurements with each hand, maximum value 30 kg if male or 20 kg if female
  3. Weight loss - Self-reported weight loss >4.5 kg (10 lbs) or >5% body weight in past 12 months
  4. Exhaustion - Two-item Center for Epidemiologic Studies Depression (CES-D) scale 1 out of 2
  5. Depression - Five-item Geriatric Depression Scale (5-GDS) 2 out of 5
  6. Low physical activity - Paffenbarger Physical Activity Index <383 kcal per week if male or < 270 kcal per week if female
  7. Cognitive impairment - Montreal Cognitive Assessment (MoCA) score <26 out of 30
Childhood retrospective circumstances questionnaire (adapted from the US Panel Study on Income Dynamics) | Baseline
  Childhood retrospective circumstances questionnaire (adapted from the US Panel Study
Weight | Baseline
  Participants change into lightweight scrub tops and bottoms, with shoes removed, to the nearest 0.1 kg using a digital calibrated floor scale
Height | Baseline
  Measured, without shoes, to the nearest 0.1 cm using a stadiometer
Body mass index (BMI) | Baseline
  Calculated as kg/m^2
Waist circumference | Baseline
  Measured in triplicate, to the nearest 0.1 cm at the umbilicus, between the last rib and the iliac crest using a fibreglass tape measure
Hip circumference | Baseline
  Measured in triplicate at the widest portion of the buttocks and hips using a fibreglass tape measure
Blood pressure | Baseline
  Systolic and diastolic blood pressures are measured in triplicate, on the non-dominant arm in a sitting position using a validated oscillometric blood pressure monitor
Pulse wave velocity | Day 1 and Day 2
  Measured on the non-dominant arm in a sitting position using a Mobil-O-Graph PWA Monitor on two consecutive days
Augmentation index | Day 1 and Day 2
  Measured on the non-dominant arm in a sitting position using a Mobil-O-Graph PWA Monitor on two consecutive days
Blood total cholesterol | Baseline
  Blood total cholesterol
Blood low-density lipoprotein cholesterol | Baseline
  Blood low-density lipoprotein cholesterol
Blood high-density lipoprotein cholesterol | Baseline
  Blood high-density lipoprotein cholesterol
Blood triglycerides | Baseline
  Blood triglycerides
Blood glucose | Baseline
  Blood glucose
Blood insulin | Baseline
  Blood insulin
Blood urea | Baseline
  Blood urea
Blood creatinine | Baseline
  Blood creatinine
Blood high sensitivity C-reactive protein | Baseline
  Blood high sensitivity C-reactive protein
Blood aspartate aminotransferase | Baseline
  Blood aspartate aminotransferase
Blood alanine aminotransferase | Baseline
  Blood alanine aminotransferase
Blood T regulatory cells | Baseline
  Blood T regulatory cells
Blood leptin | Baseline
  Blood leptin
Blood glucagon | Baseline
  Blood glucagon
Urinary melatonin | Baseline
  Urinary melatonin
Red blood cell fatty acids | Baseline
  Red blood cell fatty acids
Plasma fatty acids | Baseline
  Plasma fatty acids
Blood non-cholesterol sterols | Baseline
  Blood non-cholesterol sterols
Blood vitamin C levels | Baseline
  Blood vitamin C levels
Fractional cholesterol synthesis rate | Baseline
  Fractional cholesterol synthesis rate
Triglyceride synthesis rate | Baseline
  Triglyceride synthesis rate
Gastrointestinal microbiome | Baseline
  Microbiome 16S RNA sequencing
Physical activity level | 1 week
  Assessed using accelerometers over a period of 1 week
Muscle strength | Baseline
  Measured using a hand grip dynamometer
Cardiorespiratory fitness | Baseline
  Assessed using a metabolic cart to measure oxygen consumption (VO2; mL O2/kg body weight/minute) during a submaximal YMCA bike protocol performed to 85% of age predicted heart rate max
Functional walking ability | Baseline
  Assessed using a 5-meter gait speed test
Sleep | 1 week
  Average hours of sleep per night; measured using accelerometers over a period of 1 week
Identification and characterization of susceptibility genes for negative outcomes of lifestyle factors | Baseline
  This is meant to be achieved through a Genome Wide Association Study (GWAS) of Single Nucleotide Polymorphism (SNPs) associated with the measures of the lifestyle factors assessed in the TMPLR cohort, as listed in "outcome measures".
  Whole genome genotyping will be conducted with a state of the art genotyping array.
Identification and characterization of susceptibility genes for negative outcomes of lifestyle factors. | Baseline
  This is meant to be achieved targeted resequencing of target genes know to effect the metabolic traits assessed. This will aid the detection rare of Single Nucleotide Variations (SNVs) impacting the genes functions. Targeted re-sequencing will be conducted with a state of the art methodology.
Early life experiences by self report | Baseline
  Assessed using the childhood retrospective circumstances questionnaire (adapted from the US Panel Study on Income Dynamics
Early life experiences by maternal report | Baseline
  Assessed using a mother's questionnaire (adapted from the Nurses' Health Study)
Early life health conditions from linked administrative health records, from the Manitoba Population Healthy Research Data Repository | Baseline
  Examples of health records include: prescriptions, physician diagnoses and hospital discharge abstracts

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Study Director — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Mackay D, Mollard RC, Granger M, Bruce S, Blewett H, Carlberg J, Duhamel T, Eck P, Faucher P, Hamm NC, Khafipour E, Lix L, McMillan D, Myrie S, Ravandi A, Tangri N, Azad M, Jones PJ. The Manitoba Personalized Lifestyle Research (TMPLR) study protocol: a multicentre bidirectional observational cohort study with administrative health record linkage investigating the interactions between lifestyle and health in Manitoba, Canada. BMJ Open. 2019 Oct 10;9(10):e023318. doi: 10.1136/bmjopen-2018-023318. PMID 31604781